CLINICAL TRIAL: NCT03266367
Title: The Role of Serum Neutrophil Gelatinase Associated Lipocalin in Predicting Acute Kidney Injury in Patients With Coronary Artery Disease
Brief Title: Neutrophil Gelatinase Associated Liocalin in Predicting AKI in Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bassant Rashad, Resident Doctor, Assiut University
Other Study IDs: NGAL in AKI
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: NGAL and renal functions will be measured two hours after Percutaneous coronary intervention and two days later as a follow up
  Interventions: Diagnostic Test: Neutrophil gelatinase-associated lipocalin (NAGL)
- Healthy Group: control group
  Interventions: Diagnostic Test: Neutrophil gelatinase-associated lipocalin (NAGL)

INTERVENTIONS:
Diagnostic Test: Neutrophil gelatinase-associated lipocalin (NAGL) — Serum level of Neutrophil gelatinase-associated lipocalin (NAGL) using the enzyme linked immunosorbent assay kits (ELISA)

SUMMARY:
The aim of this work is to assess the clinical significance of serum levels of neutrophil gelatinase-associated lipocalin (NGAL) to predict AKI in patients exposed to PCI.

DETAILED DESCRIPTION:
ST-elevated myocardial infarction(STEMI) patients are at a particularly high risk of acute kidney injury (AKI) because of the complexity of hemodynamic disorders and adverse effects associated with the use of radiopaque diagnostic and treatment methods (Smirnov AV.et al.,2009) With wide application of percutaneous coronary intervention (PCI) technology in patients with coronary artery disease (CAD), contrast-induced acute kidney injury (CI-AKI) has become a serious complication and is the third leading cause of AKI in hospitalized patients.(Gleeson.et al. 2004)

To date,AKI diagnosis has been limited to observation of increasing levels of serum creatinine,decrease in urine output,and alterations in urinary chemistry (Bellomo.et al.2004;Mehta.et al. 2007) Nevertheless,serum creatinine levels do not increase significantly until renal function has decreased to 50% in addition,the level of serum creatinine may be affected by the patient's muscle mass,catabolic state,protein intake,weight,sex and tubular secretion of creatinine.Therefore,applying serum creatinine as a biomarker for diagnosing AKI may result in the loss of valuable time (Mishra.et al.2005;Sirota.et al.2011)

Neutrophil Gelatinase-associated lipocalin(NGAL) belongs to the lipocalin family and is produced predominantly by the liver and white blood cells(Hvidberg.et al.,2005).

A small polypeptide, neutrophil gelatinase-associated lipocalin (NGAL), is one of the most promising and best-studied AKI biomarkers (Mishra.et al.,2003; Devarajan.et al 2003) The expression of NGAL was predominantly in proliferating and regenerating tubular epithelial cells, which suggested a role in repair. (Mori.et al.2005) The majority of NGAL, secreted by injured renal tubule epithelial cells, is in a 25kDa monomeric form. In contrast, neutrophils have been claimed to release NGAL primarily as a 45kDa homodimer, i.e. two NGAL monomers linked by a disulfide bridge. It also exists as a 135-kDa heterodimer, covalently conjugated with gelatinase (Cai.et al.2010) NGAL is easily detected in blood and urine due to its small size and resistance to degradation. It can be measured non-invasively using routine laboratory analysers as well as some point of care devices. Furthermore, NGAL concentration in both urine and plasma rises rapidly in a dose-dependent manner that is proportional to the degree of acute kidney damage (Haase-Fielitz.et al.2009)

NGAL has previously been termed the 'troponin-like' biomarker to detect subclinical AKI even in the absence of diagnostic increases in SCr (Devarajan.,2010;Haase,et al.2011) Additionally, NGAL has been reported to be predictive 48 h prior to the actual time of injury; therefore, renal replacement therapy can be planned earlier(Cruz,et al.2010)

ELIGIBILITY:
Inclusion Criteria:

* patients exposed to percutaneous coronary intervention

Exclusion Criteria:

* 1.Diabetes mellitus 2.Liver disease 3.Chronic Kidney Disease 4.Renal Replacement Therapy 5.Previous kidney transplant 6.Chronic infection

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all male and female patients with coronary artery disease who are recently exposed to PCI (20_70 years old )
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
The rise of NGAL in AKI after PCI before rise of renal function | 2 days

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Result] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Result] Mishra J, Dent C, Tarabishi R, Mitsnefes MM, Ma Q, Kelly C, Ruff SM, Zahedi K, Shao M, Bean J, Mori K, Barasch J, Devarajan P. Neutrophil gelatinase-associated lipocalin (NGAL) as a biomarker for acute renal injury after cardiac surgery. Lancet. 2005 Apr 2-8;365(9466):1231-8. doi: 10.1016/S0140-6736(05)74811-X. PMID 15811456
- [Result] Hvidberg V, Jacobsen C, Strong RK, Cowland JB, Moestrup SK, Borregaard N. The endocytic receptor megalin binds the iron transporting neutrophil-gelatinase-associated lipocalin with high affinity and mediates its cellular uptake. FEBS Lett. 2005 Jan 31;579(3):773-7. doi: 10.1016/j.febslet.2004.12.031. PMID 15670845
- [Result] Mishra J, Ma Q, Prada A, Mitsnefes M, Zahedi K, Yang J, Barasch J, Devarajan P. Identification of neutrophil gelatinase-associated lipocalin as a novel early urinary biomarker for ischemic renal injury. J Am Soc Nephrol. 2003 Oct;14(10):2534-43. doi: 10.1097/01.asn.0000088027.54400.c6. PMID 14514731
- [Result] Devarajan P, Mishra J, Supavekin S, Patterson LT, Steven Potter S. Gene expression in early ischemic renal injury: clues towards pathogenesis, biomarker discovery, and novel therapeutics. Mol Genet Metab. 2003 Dec;80(4):365-76. doi: 10.1016/j.ymgme.2003.09.012. PMID 14654349
- [Result] Mori K, Lee HT, Rapoport D, Drexler IR, Foster K, Yang J, Schmidt-Ott KM, Chen X, Li JY, Weiss S, Mishra J, Cheema FH, Markowitz G, Suganami T, Sawai K, Mukoyama M, Kunis C, D'Agati V, Devarajan P, Barasch J. Endocytic delivery of lipocalin-siderophore-iron complex rescues the kidney from ischemia-reperfusion injury. J Clin Invest. 2005 Mar;115(3):610-21. doi: 10.1172/JCI23056. PMID 15711640
- [Result] Cai L, Rubin J, Han W, Venge P, Xu S. The origin of multiple molecular forms in urine of HNL/NGAL. Clin J Am Soc Nephrol. 2010 Dec;5(12):2229-35. doi: 10.2215/CJN.00980110. Epub 2010 Sep 9. PMID 20829422
- [Result] Haase-Fielitz A, Bellomo R, Devarajan P, Bennett M, Story D, Matalanis G, Frei U, Dragun D, Haase M. The predictive performance of plasma neutrophil gelatinase-associated lipocalin (NGAL) increases with grade of acute kidney injury. Nephrol Dial Transplant. 2009 Nov;24(11):3349-54. doi: 10.1093/ndt/gfp234. Epub 2009 May 27. PMID 19474273
- [Result] Haase M, Devarajan P, Haase-Fielitz A, Bellomo R, Cruz DN, Wagener G, Krawczeski CD, Koyner JL, Murray P, Zappitelli M, Goldstein SL, Makris K, Ronco C, Martensson J, Martling CR, Venge P, Siew E, Ware LB, Ikizler TA, Mertens PR. The outcome of neutrophil gelatinase-associated lipocalin-positive subclinical acute kidney injury: a multicenter pooled analysis of prospective studies. J Am Coll Cardiol. 2011 Apr 26;57(17):1752-61. doi: 10.1016/j.jacc.2010.11.051. PMID 21511111
- [Result] Cruz DN, de Cal M, Garzotto F, Perazella MA, Lentini P, Corradi V, Piccinni P, Ronco C. Plasma neutrophil gelatinase-associated lipocalin is an early biomarker for acute kidney injury in an adult ICU population. Intensive Care Med. 2010 Mar;36(3):444-51. doi: 10.1007/s00134-009-1711-1. Epub 2009 Dec 3. PMID 19956925